CLINICAL TRIAL: NCT03568006
Title: Effectiveness of Passive Mobilization of Glenohumeral Joint in Patients With Subacromial Syndrome: a Randomized Controlled Trial
Brief Title: Effectiveness of Passive Mobilization in Patients With Subacromial Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Collaborators: Montpellier Clinic (Unknown)
Responsible Party: Principal Investigator, Pablo Herrero Gallego, Dr. Pablo Herrero, PT, PhD. Head of iPhysio Research Group., Universidad San Jorge
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TM_AJ
Record Dates: First submitted 2018-06-12; First posted 2018-06-26 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Subacromial Impingement
Keywords: subacromial impingement; pain; shoulder; passive mobilization
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: It is not possible to mask physiotherapists and patients, so the only masking will be for researchers and evaluators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention will consist of passive joint mobilization (caudal and dorsal gliding) grade II in the glenohumeral joint.
  Besides, participants will receive a standardized treatment consisting of infrared rays, a program of therapeutic exercises and indications to improve their postural hygiene.
  Interventions: Other: Specific passive mobilization; Other: Standardized treatment (standard protocol)
- Control (Active Comparator): Control treatment will consist of a standardized treatment consisting of infrared rays, a program of therapeutic exercises and indications to improve their postural hygiene.
  Interventions: Other: Standardized treatment (standard protocol)

INTERVENTIONS:
Other: Specific passive mobilization — Specific passive mobilizations for the shoulder
  Arms: Intervention
Other: Standardized treatment (standard protocol) — Infrared rays, a program of therapeutic exercises and indications to improve their postural hygiene

SUMMARY:
From a biomechanical point of view, subacromial syndrome causes an increment in the anterior and superior translation of the humeral head, which increases compression in the adjacent tissues of the subacromial space, aggravating the symptoms of the patients. Conservative treatments are the first option for subacromial syndrome management, despite the fact that there is limited evidence about its effectiveness, due to the lack of experimental studies.

The aim of this study is to evaluate the effectiveness of a passive joint mobilization (caudal and dorsal gliding) grade II in the glenohumeral joint, within a multimodal approach to reduce pain and improve the range of motion in patients with subacromial syndrome.

DETAILED DESCRIPTION:
Subacromial syndrome, also known as subacromial impingement, is the most frequent disorder in the shoulder joint. It has a multifactorial origin and represents a wide spectrum of pathologies. Its main consequences are pain and loss of function in the glenohumeral joint. From a biomechanical point of view, subacromial syndrome causes an increment in the anterior and superior translation of the humeral head, which increases compression in the adjacent tissues of the subacromial space, aggravating the symptoms of the patients. Conservative treatments are the first option for subacromial syndrome management, despite the fact that there is limited evidence about its effectiveness, due to the lack of experimental studies.

The aim of this study is to evaluate the effectiveness of a passive joint mobilization (caudal and dorsal gliding) grade II in the glenohumeral joint, within a multimodal approach to reduce pain and improve the range of motion in patients with subacromial syndrome. To this end, a randomized clinical trial will be carried out in the Montpellier Clinic in Zaragoza. Twenty-two patients will be recruited and randomly assigned to one of the two groups (intervention and control). Both groups will receive a standardized treatment consisting of: 10 sessions of infrared rays, and a program of therapeutic exercises and indications to improve their postural hygiene. In addition, the intervention group will receive a passive joint mobilization in the glenohumeral joint of 5 minutes. Pain intensity, range of motion and functionality of the glenohumeral joint will be measured in the first session before any treatment and in the tenth session after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subacromial syndrome
* Pain at rest, which increases when doing active movements
* Neer´s impingement test positive
* Hawkins Kennedy test positive
* Pain lasting more than one month
* Anteriorization of humeral head
* Full capacity (physical and cognitive) to participate in the study and give consent.

Exclusion Criteria:

* Infiltrations during the previous six months
* Traumatic origin of pain
* Complete tear of any rotator cuff tendon
* Bilateral pain
* Previous surgical intervention in the affected shoulder
* Patients planning to start with other treatments during the clinical trial.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change between baseline (immediately before intervention) and post intervention (2 weeks).
  10 centimetres Visual Analogue Scale. 0 is no pain, whilst 10 is maximum intolerable pain

SECONDARY OUTCOMES:
Active range of motion | Change between baseline (immediately before intervention) and post intervention (2 weeks).
  Measurement of active range of motion for the different shoulder movements (abduction from 0 to 150º, flexion from 0 to 180º, extension from 0 to 60º, lateral rotation from 0 to 90º, internal rotation from o to 70º)
Constant Score | Change between baseline (immediately before intervention) and post intervention (2 weeks).
  Scale to measure shoulder function, ranging from 0 to 100. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient.[1] The Constant score was introduced to determine the functionality after the treatment of a shoulder injury. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.

CONTACTS AND LOCATIONS:
Locations (1):
- San Jorge University, Villanueva de Gállego, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No